CLINICAL TRIAL: NCT04817293
Title: Coordinated Research on Prolonged Symptoms and Reasons for Consultation in Town Medicine Associated With SARS-COV-2 Infection: a Transversal Study in Town in the Hauts de France Region
Brief Title: Prolonged Symptoms and Reasons for Consultation in Town Medicine Associated With COVID-19 Infection in the Hauts de France Region
Acronym: COCO_Vi_LATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH_2021_01
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive
  Interventions: Other: Questionnaire; Other: medical consultation
- COVID-19 negative
  Interventions: Other: Questionnaire; Other: medical consultation

INTERVENTIONS:
Other: Questionnaire — Questionnaire SSD-12 and EQ5D5L
Other: medical consultation — Medical consultation during the visit with data collection

SUMMARY:
Several publications document the occurrence of prolonged or late-onset symptoms beyond 3 weeks after the first clinical manifestations of SARS-COV2 infection. These manifestations may be related to thromboembolic or inflammatory events or other mechanisms that are not yet well understood. The psychosomatic origin secondary to psychiatric disorders prior to the infection or in reaction to it is also to be evoked. The identification of the clinical manifestations observed, and their clinical and paraclinical evolution are essential to better understand the natural evolution of COVID-19, to specify the physiopathological mechanisms and to identify potential avenues of management for the patients. In addition, the impact of COVID-19 infection on primary care visits is not known. In general practice, these patients benefit from explorations and even diagnoses that may explain the persistence of symptoms (autoimmune diseases, thrombosis, somatoform disorders, hyperventilation syndrome, etc.).

The objective of the COCO_Vi_LATE project is to carry out a cross-sectional study of patients presenting persistent and/or recurrent symptoms after an infection with SARS-COV-2 who will be compared to individuals with a short form of infection with COVID-19

ELIGIBILITY:
Inclusion Criteria:

A- For COVID cases:

1. Consultation in a city doctor's office
2. Positive SARS-CoV-2 RT-PCR result OR positive SARS-CoV-2 serology
3. Patient symptomatic or not

Definition of symptomatic :

1. Anosmia
2. OR CT scan suggestive of COVID 19
3. OR ≥ 2 symptoms contemporaneous with virologic sampling among: asthenia, cough, dyspnea, fever, myalgias, dysgeusia, diarrhea AND not present previously at diagnosis

B-. For NON COVID cases:

1. Consultation in a city doctor's office
2. No known COVID+ serology
3. No known RT- PCR SARS-CoV-2
4. No clinical suspicion of COVID-19 infection

Exclusion Criteria:

1. Minor patient
2. Refusal to participate
3. Patient under protection
4. Patient requiring hospitalization for COVID-19 (excluding non-emergency hospitalization)
5. Patient consulted for the following reason only: treatment monitoring, treatment renewal or certificate, hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: he study population consisted of patients with COVID-19 infection and patients without COVID-19 infection consulting their general practitioner during the study inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
To compare the reasons for consultation between patients with a history of Covid 19 and those who have not been infected with SARS-CoV-2. | At day 1
  The judgement criterion will be the reasons for consultation standardized with the CISP-2 classification (International Classification of Primary Care).

SECONDARY OUTCOMES:
To Assess the presence of somatoform disorders between COVID-19 and non-COVID-19 patients. | At day 1
  The assessment will be done using the international SSD-12 scale (Symptom Disorder-B Criteria Scale). The SSD-12 is composed of 12 items; each of the three psychological subcriteria is measured by four items (cognitive aspects; affective aspects; behavioral aspects).
To compare the quality of life of COVID-19 patients with that of non-COVID-19 patients. | At day 1
  The EQ-5D-5L scale is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier ROBINEAU, MD, Principal Investigator — CH TOURCOING; Sophie PANAGET, MD, Principal Investigator — CHRU LILLE
Locations (1):
- CH Tourcoing, Tourcoing, France

IPD SHARING:
Plan to Share IPD: No